CLINICAL TRIAL: NCT03106662
Title: Mesenchymal Stem Cell Infusion in Haploidentical Hematopoietic Stem Cell Transplantation in Patients With Hematological Malignancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Onder Arslan, MD, Department of Hematology, Clinical Professor, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213S196
Record Dates: First submitted 2015-11-13; First posted 2017-04-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Mesenchymal stem cell; haploidentical hematopoietic stem cell transplantation; graft-versus-host disease; engraftment
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal Stem Cell in Haplo-SCT (Experimental): After preferred conditioning regimen for the patient, cyclophosphamide 50 mg/kg/day will be administered at +3 and +4 post transplant day. At +6 post transplant day, 2-8x10^8 cell/kg mesenchymal stem cells will be infused.
  Interventions: Biological: mesenchymal stem cells; Drug: cyclophosphamide administration

INTERVENTIONS:
Biological: mesenchymal stem cells — After preferred conditioning regimen for the patient, cyclophosphamide 50 mg/kg/day will be administered at +3 and +4 post transplant day. At +6 post transplant day, 2-8x10^8 cell/kg mesenchymal stem cells will be infused.
Drug: cyclophosphamide administration — After preferred conditioning regimen for the patient, cyclophosphamide 50 mg/kg/day will be administered at +3 and +4 post transplant day.

SUMMARY:
Mesenchymal stem cells (MSCs) have been used in the treatment and prevention of graft-versus host disease (GVHD). In this study the investigators aim to present the efficacy of mesenchymal stem cells in graft versus host disease prophylaxis and effect of engraftment in haploidentical recipients. Forty patients aged older than 18 who have indications for haploidentical hematopoietic stem cell transplantation will be included to the study. MSCs will be isolated from donor bone marrows and infused to the patient after conditioning regimen on day +6. If the haploidentical transplantation results improve with MSCs treatment it would be possible to ameliorate the problem of HLA-matched donor paucity in Turkey and prefer haploidentical donors.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs) have been utilized in the treatment and prevention of graft-versus-host disease(GVHD) after allogeneic hematopoietic stem cell transplantation (alloSCT). However, studies on MSC use in alloSCT from haploidentical donors (haploSCT) have been limited.

In this study, the investigators aim 1) to evaluate MSCs' efficacy in GVHD prophylaxis and effect on engraftment of the haploidentical graft, 2) to improve the success rate of haploSCT by further decreasing GVHD incidence and graft failure rate. With higher haploSCT success rates, haploidentical donors would be important alternative graft sources in patients without HLA-matched donors.

Forty patients who present to Ankara University, School of Medicine, Division of Hematology with hematological malignancies and have indications for haploSCT will be included in the study after informed consent is obtained. MSCs will be procured and isolated from donor bone marrows. MSCs will be isolated, cultured, and stored in the good manufacturing practice (GMP) laboratory in Ankara University Stem Cell Institute. Donor bone marrow will be harvested, four to six weeks prior to transplantation, for MSC isolation and culture. Patients will receive either an ablative or non-ablative induction regimen based on their age, diagnosis, and the disease status at the time of transplantation. Donor bone marrow will be harvested a second time on the day of transplantation and the procured bone marrow graft will be infused to the patient the same day. GVHD prophylaxis will include post-transplantation cyclophosphamide (Cy) on days +3 and +4 (50 mg/kg/day), tacrolimus, and mycophenolate mofetil. Stored MSCs will be infused to the patient on day +6. The endpoints include graft failure rate, GVHD incidence, transplant-related mortality, disease-free survival, and overall survival.

The investigators aim to evaluate the utility of MSCs in improving haploSCT results and to enhance the reliability and success of haploSCT. Successful transplants from haploidentical donors would ameliorate the problem of matched donor paucity in countries with a limited number of hematopoietic stem cell donors, such as Turkey, and would establish haploidentical donors an alternative donor source for patients without matched donors in Turkey. As haploidentical donors may be parents or children, rapid and easy access to donors would decrease wait times for alloSCT. Moreover, national current account deficit may be reduced through using grafts obtained from haploidentical donors residing in Turkey instead of grafts from foreign stem cell/umbilical cord banks.

In this project, the investigators seek to develop clinical therapy applications in concordant with the ambition of "renewal and repair of human cells, tissues, and organs through cellular therapy and cellular products" that is included in the The Scientific and Technological Research Council of Turkey 1003 Call for Projects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with haematological malignancy
* Indication of haploidentical hematopoietic stem cell transplantation
* No restrictions for transplantation

Exclusion Criteria:

* Any restriction for transplantation
* No indication of haploidentical hematopoietic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-10; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Effect of mesenchymal stem cells on overall survival in haploidentical stem cell transplantation | 36 months

SECONDARY OUTCOMES:
Effect of mesenchymal stem cells on graft versus host disease incidence in haploidentical stem cell transplantation | 36 months
Effect of mesenchymal stem cells on graft failure incidence in haploidentical stem cell transplantation | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School of Medicine Department of Hematology, Ankara, Turkey (Türkiye)